CLINICAL TRIAL: NCT00666003
Title: Hemodynamic Assessment Comparison Between Arterial Pressure Cardiac Output Monitor and Crit Line Utilized During Renal Replacement Therapy
Brief Title: Hemodynamic Assessment APCO Monitor vs Crit Line for Renal Replacement Rx
Acronym: APCOvC-Line
Status: Completed | Type: Observational
Sponsor: Baystate Medical Center (Other)
Responsible Party: Patrick T. Mailloux, DO, Baystate Medical Cetner
Other Study IDs: IRB07-120
Record Dates: First submitted 2008-04-23; First posted 2008-04-24 (Estimated); Last update posted 2011-02-08 (Estimated); Status verified 2011-02

CONDITIONS: Renal Failure; Hemodynamics
Keywords: Hemodynamics
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Fluid and volume management are a challenging part of critical care and the difficulties increase in the face of renal failure. Utilizing the Crit-Line to monitor blood volume changes in conjunction with arterial pressure cardiac output monitoring may lead to better understanding of the impact fluid removal during dialysis has on hemodynamics.

DETAILED DESCRIPTION:
Patients in an ICU often require large amounts of IV fluid to maintain adequate cardiac function. In patients with renal failure, the ability to gauge adequacy of circulating blood volume based on urine output is obviously lacking. The FDA approved devices called Flotrac/Vigileo and Crit-Line are used in this setting to determine adequacy of fluid resuscitation. This study proposes to use the data collected in a retrospective manner to determine if correlation of the various measured parameters can serve as a predictor of hemodynamic status.

ELIGIBILITY:
Inclusion Criteria:

* Indwelling arterial catheter
* Require dialysis
* CVP in place
* Use of Crit-Line and Flotrak device

Exclusion Criteria:

* Aortic Regurgitation
* Use of an intra-aortic balloon pump
* Weight less than 90 lbs
* Cardiac arrhythmias

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Renal Failure Patients in the ICU
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2008-04; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Mailloux, D.O., Principal Investigator — Baystate Medical Center
Locations (1):
- Baystate Medical Center, Springfield, Massachusetts, United States